CLINICAL TRIAL: NCT02101554
Title: AN OPEN-LABEL STUDY TO EVALUATE THE SAFETY AND PHARMACOKINETICS OF PF-06412528 IN CHILDREN 7-17 YEARS FOR THE TREATMENT OF MODERATE-TO-SEVERE PAIN
Brief Title: Safety and Pharmacokinetic Study of EMBEDA in Children Ages 7-17 With Pain
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Pfizer released from post-marketing commitment and study terminated because too few patients in the age group; not because of efficacy or safety issues.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: B4541006; EMBEDA (Other: Alias Study Number)
Record Dates: First submitted 2014-03-05; First posted 2014-04-02 (Estimated); Results first posted 2020-07-10 (Actual); Last update posted 2020-07-10 (Actual); Status verified 2020-06

CONDITIONS: Moderate-severe Pain
Keywords: Pediatric; pain indication; controlled release morphine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Embeda (Experimental): One arm, open label, active
  Interventions: Drug: Ages 7-11; Drug: ages 12-17

INTERVENTIONS:
Drug: Ages 7-11 — Oral/Capsule, once per day or twice per day dosing; Treatment duration consists of a 1 to 4 week Conversion/Titration Phase leading to a 2 to 6 week Maintenance Treatment duration.
Drug: ages 12-17 — Oral/Capsule, once per day or twice per day dosing; Treatment duration consists of a 1 to 4 week Conversion/Titration Phase leading to a 2 to 6 week Maintenance Treatment duration.

SUMMARY:
Safety and pharmacokinetics of an abuse-deterrent, extended-release formulation of morphine sulfate with a sequestered naltrexone core in children 7-17 with moderate-severe pain.

DETAILED DESCRIPTION:
Subjects, once stabilized to Embeda, need only complete a minimum of 2 of the 6 week study duration to satisfy the PK endpoint. A safety follow-up visit is required at 1 week post-last dose.

ELIGIBILITY:
Inclusion Criteria:

* Children 7-17 with moderate to severe pain requiring around the clock treatment with an opioid analgesic.
* Be an experienced opioid user, defined as any subject treated with opioid therapy, equivalent or equal to >20 mg per day of morphine, for a period of 3 consecutive days immediately prior to first day of dosing.

Exclusion Criteria:

* Columbia-Suicide Severity Rating Scale (C-SSRS) for suicidal ideation and behavior in past year.
* Hypersensitivity to morphine, naltrexone.
* A life expectancy (assessed by investigator) of less than 6 months or is no longer capable of taking medication orally.
* Undergone surgery within 3 days prior to the first day of dosing.

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 19 (Actual)
Dates: Start 2015-04-24 (Actual); Primary Completion 2019-06-26 (Actual); Study Completion 2019-06-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (19):
- United States (19):
  - Gottschalk Medical Plaza, Irvine, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - The University of California, Irvine Health - Medical Specialties, Orange, California
  - UCI Medical Center- Outpatient Pharmacy, Orange, California
  - University of California, Irvine Health-Inpatient Pharmacy, Orange, California
  - University of California, Irvine Health-Medical Specialties, Orange, California
  - Holtz Children Hospital/Jackson Memorial Hospital, Miami, Florida
  - Jackson Memorial Hospital - Pharmacy Department Basement West, Miami, Florida
  - Sylvester Comprehensive Cancer Center-Alex's Place, Miami, Florida
  - University of Miami / Jackson Memorial Hospital, Miami, Florida
  - Nicklaus Children's Hospital, Miami, Florida
  - Veritas Research Corp., Miami Lakes, Florida
  - University of Illinois at Chicago Clinical Research Center, Chicago, Illinois
  - University of Illinois at the Med Center, University of Illinois, Chicago, Illinois
  - University of Illinois Hospital and Health Sciences System, Chicago, Illinois
  - East Carolina University Brody School of Medicine(ECU), Greenville, North Carolina
  - Leo Jenkins Cancer Center Pharmacy Attn: Rebecca Turnage, Greenville, North Carolina
  - Primary Children's Hospital Outpatient Services, Salt Lake City, Utah
  - Primary Children's Hospital, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B4541006&StudyName=Safety%20and%20Pharmacokinetic%20Study%20of%20EMBEDA%20in%20Children%20Ages%207-17%20with%20Chronic%20Pain

RESULTS

PARTICIPANT FLOW:
Groups:
- PF-06412528 <=20 mg: Participants were converted from their pre-study standard of care opioid analgesic to PF-06412528; PF-06412528 oral dose was titrated and stabilized to less than or equal to (<=) 20 milligram (mg) daily, up to a maximum of 4 weeks. Participants continued to receive stabilized PF-06412528 <=20 mg oral daily dose up to a maximum of additional 6 weeks.
- PF-06412528 >20-40 mg: Participants were converted from their pre-study standard of care opioid analgesic to PF-06412528; PF-06412528 oral dose was titrated and stabilized to greater than (>) 20 mg to 40 mg daily, up to a maximum of 4 weeks. Participants continued to receive stabilized PF-06412528 >20 mg to 40 mg oral daily dose up to a maximum of additional 6 weeks.
- PF-06412528 >40-80 mg: Participants were converted from their pre-study standard of care opioid analgesic to PF-06412528; PF-06412528 oral dose was titrated and stabilized to >40 mg to 80 mg daily, up to a maximum of 4 weeks. Participants continued to receive stabilized PF-06412528 >40 mg to 80 mg oral daily dose up to a maximum of additional 6 weeks.
Period: Overall Study
Arm/Group | PF-06412528 <=20 mg | PF-06412528 >20-40 mg | PF-06412528 >40-80 mg
Started | 6 | 10 | 3
Completed | 3 | 5 | 2
Not Completed | 3 | 5 | 1
Not completed — Protocol Violation | 0 | 1 | 0
Not completed — Insufficient Clinical Response | 0 | 2 | 0
Not completed — Adverse Event | 2 | 1 | 1
Not completed — Lost to Follow-up | 0 | 1 | 0
Not completed — Withdrawl by Parents/Guardians | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety analysis population included all participants who received at least 1 dose of PF-06412528.
Groups:
- Total: Total of all reporting groups
Arm/Group | PF-06412528 <=20 mg | PF-06412528 >20-40 mg | PF-06412528 >40-80 mg | Total
Number analyzed (Participants) | 6 | 10 | 3 | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.3 (2.34) | 15.0 (1.33) | 15.3 (1.53) | 14.8 (1.68)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 7 | 3 | 13
  Male | 3 | 3 | 0 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 4 | 0 | 8
  Not Hispanic or Latino | 2 | 6 | 3 | 11
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 2 | 2 | 2 | 6
  White | 3 | 7 | 1 | 11
  More than one race | 1 | 1 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs): Week 1 to Week 4
Description: An AE was any untoward medical occurrence in a participant who received study treatment without regard to possibility of causal relationship. SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death, initial or prolonged inpatient hospitalization, life-threatening experience (immediate risk of dying), persistent or significant disability or incapacity, congenital anomaly. A treatment emergent AE was defined as an event that emerged during the treatment period that was absent before treatment, or worsened during the treatment period relative to the pretreatment state. AEs included both serious and non-serious adverse events.
Time Frame: Week 1 to Week 4
Population: Analysis population included all participants who were screened and had received at least 1 dose of PF-06412528 from Week 1 to Week 4.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-06412528 <=20 mg | PF-06412528 >20-40 mg | PF-06412528 >40-80 mg
Number analyzed (Participants) | 6 | 10 | 3
Participants
  AEs | 4 | 9 | 3
  SAEs | 1 | 1 | 1

2. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs): Week 5 to Week 10
Description: as for outcome 1
Time Frame: Week 5 to Week 10
Population: Analysis population included all participants who were screened and had received at least 1 dose of PF-06412528 from Week 5 to Week 10.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-06412528 <=20 mg | PF-06412528 >20-40 mg | PF-06412528 >40-80 mg
Number analyzed (Participants) | 4 | 8 | 2
Participants
  AEs | 3 | 7 | 2
  SAEs | 1 | 2 | 1

3. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events According to Severity: Week 1 to Week 4
Description: An adverse event was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. AE was assessed according to severity; mild (does not interfere with participant's usual function), moderate (interferes to some extent with participant's usual function) and severe (interferes significantly with participant's usual function).A treatment emergent AE was defined as an event that emerged during the treatment period that was absent before treatment, or worsened during the treatment period relative to the pretreatment state. AEs included both serious and non-serious adverse events.
Time Frame: Week 1 to Week 4
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | PF-06412528 <=20 mg | PF-06412528 >20-40 mg | PF-06412528 >40-80 mg
Number analyzed (Participants) | 6 | 10 | 3
Participants
  Mild | 1 | 4 | 2
  Moderate | 0 | 3 | 0
  Severe | 3 | 2 | 1

4. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events According to Severity: Week 5 to Week 10
Description: An adverse event was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. AE was assessed according to severity; mild (does not interfere with participant's usual function), moderate (interferes to some extent with participant's usual function) and severe (interferes significantly with participant's usual function). A treatment emergent AE was defined as an event that emerged during the treatment period that was absent before treatment, or worsened during the treatment period relative to the pretreatment state. AEs included both serious and non-serious adverse events.
Time Frame: Week 5 to Week 10
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | PF-06412528 <=20 mg | PF-06412528 >20-40 mg | PF-06412528 >40-80 mg
Number analyzed (Participants) | 4 | 8 | 2
Participants
  Mild | 1 | 3 | 0
  Moderate | 1 | 2 | 0
  Severe | 1 | 2 | 2

5. Primary Outcome: Number of Participants With Treatment Emergent Treatment Related Adverse Events: Week 1 to Week 4
Description: An AE was any untoward medical occurrence attributed to study drug in a participant who received study drug. A treatment emergent AE was defined as an event that emerged during the treatment period that was absent before treatment, or worsened during the treatment period relative to the pretreatment state. Relatedness to PF-06412528 was assessed by the investigator.
Time Frame: Week 1 to Week 4
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | PF-06412528 <=20 mg | PF-06412528 >20-40 mg | PF-06412528 >40-80 mg
Number analyzed (Participants) | 6 | 10 | 3
Participants | 2 | 4 | 0

6. Primary Outcome: Number of Participants With Treatment Emergent Treatment Related Adverse Events: Week 5 to Week 10
Description: as for outcome 5
Time Frame: Week 5 to Week 10
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | PF-06412528 <=20 mg | PF-06412528 >20-40 mg | PF-06412528 >40-80 mg
Number analyzed (Participants) | 4 | 8 | 2
Participants | 2 | 4 | 1

7. Primary Outcome: Number of Participants With Clinical Opiate Withdrawal Scale (COWS) at Screening Before Day 1
Description: COWS is a clinician-administered instrument, to assess participants' clinical opiate withdrawal level. The scale ranges from 0 (none symptoms) to 48 (severe symptoms), higher score = more severe withdrawal. Scores category: 0 to 4 = none to minimal, 5 to 12 = mild, 13 to 24 = moderate, 25 to 36 = moderately severe withdrawal and 37 to 48 = severe withdrawal. Participants experiencing a COWS score greater than equal to (>=) 13 is treated for opiate withdrawal signs and symptoms according to the investigator's medical judgment. In this outcome measure, participants as per COWS score categories are reported. Only those COWS categories are presented which had at least 1 participant for any reporting arm.
Time Frame: At Screening (2 weeks before Day 1 of study)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | PF-06412528 <=20 mg | PF-06412528 >20-40 mg | PF-06412528 >40-80 mg
Number analyzed (Participants) | 6 | 10 | 3
Participants
  COWS Score < 5 | 6 | 9 | 3
  Mild (COWS Score 5-12) | 0 | 1 | 0

8. Primary Outcome: Number of Participants With Clinical Opiate Withdrawal Scale (COWS) at Day 1
Description: as for outcome 7
Time Frame: Day 1 (Pre-dose)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | PF-06412528 <=20 mg | PF-06412528 >20-40 mg | PF-06412528 >40-80 mg
Number analyzed (Participants) | 6 | 10 | 3
Participants
  COWS Score < 5 | 6 | 9 | 3
  Mild (COWS Score 5-12) | 0 | 1 | 0

9. Primary Outcome: Number of Participants With Clinical Opiate Withdrawal Scale (COWS) at Week 1
Description: as for outcome 7
Time Frame: Week 1
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | PF-06412528 <=20 mg | PF-06412528 >20-40 mg | PF-06412528 >40-80 mg
Number analyzed (Participants) | 6 | 10 | 3
Participants
  COWS Score < 5 | 6 | 8 | 3
  Mild (COWS Score 5-12) | 0 | 1 | 0
  Missing | 0 | 1 | 0

10. Primary Outcome: Number of Participants With Clinical Opiate Withdrawal Scale (COWS) at Week 2
Description: as for outcome 7
Time Frame: Week 2
Population: Analysis population included all participants who were screened and had received at least 1 dose of PF-06412528 from Week 1 to Week 4. Overall number of participants analyzed=0 for arm PF-06412528 >40-80 mg as no participants were evaluable for this outcome measure at Week 2.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-06412528 <=20 mg | PF-06412528 >20-40 mg | PF-06412528 >40-80 mg
Number analyzed (Participants) | 6 | 10 | 0
Participants
  COWS Score < 5 | 1 | 9 |
  Missing | 5 | 1 |

11. Primary Outcome: Number of Participants With Clinical Opiate Withdrawal Scale (COWS) at Week 3
Description: as for outcome 7
Time Frame: Week 3
Population: Analysis population: all participants who were screened and had received at least 1 dose of PF-06412528 from Week 1-4. Overall number of participants analyzed=0 for arm PF-06412528 >40-80 mg as no participants were evaluable for this outcome measure at Week 3.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-06412528 <=20 mg | PF-06412528 >20-40 mg | PF-06412528 >40-80 mg
Number analyzed (Participants) | 6 | 10 | 0
Participants
  COWS Score <5 | 1 | 3 |
  Missing | 5 | 7 |

12. Primary Outcome: Number of Participants With Clinical Opiate Withdrawal Scale (COWS) at Week 4
Description: as for outcome 7
Time Frame: Week 4
Population: Analysis population: all participants who were screened and received at least 1 dose of PF-06412528 from Week 1-4. Overall number of participants analyzed=0 for arm PF-06412528 <=20 mg and PF-06412528 >40-80 mg as no participants were evaluable for this outcome measure at Week 4.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-06412528 <=20 mg | PF-06412528 >20-40 mg | PF-06412528 >40-80 mg
Number analyzed (Participants) | 0 | 10 | 0
Participants
  COWS Score <5 |  | 2 |
  Missing |  | 8 |

13. Primary Outcome: Number of Participants With Clinical Opiate Withdrawal Scale (COWS) at Early Termination Before Week 4
Description: as for outcome 7
Time Frame: Early Termination before Week 4 (anytime between Week 1 to Week 4)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | PF-06412528 <=20 mg | PF-06412528 >20-40 mg | PF-06412528 >40-80 mg
Number analyzed (Participants) | 6 | 10 | 3
Participants
  COWS Score <5 | 2 | 2 | 1
  Missing | 4 | 8 | 2

14. Primary Outcome: Number of Participants With Clinical Opiate Withdrawal Scale (COWS) at Screening on Week 5
Description: as for outcome 7
Time Frame: Screening before treatment started at Week 5
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | PF-06412528 <=20 mg | PF-06412528 >20-40 mg | PF-06412528 >40-80 mg
Number analyzed (Participants) | 4 | 8 | 2
Participants | 4 | 8 | 2

15. Primary Outcome: Number of Participants With Clinical Opiate Withdrawal Scale (COWS) at Day 1 of Week 5
Description: as for outcome 7
Time Frame: Day 1 of Week 5
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | PF-06412528 <=20 mg | PF-06412528 >20-40 mg | PF-06412528 >40-80 mg
Number analyzed (Participants) | 4 | 8 | 2
Participants
  COWS Score <5 | 4 | 7 | 2
  Mild (COWS Score 5-12) | 0 | 1 | 0

16. Primary Outcome: Number of Participants With Clinical Opiate Withdrawal Scale (COWS) at Week 6
Description: as for outcome 7
Time Frame: Week 6
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | PF-06412528 <=20 mg | PF-06412528 >20-40 mg | PF-06412528 >40-80 mg
Number analyzed (Participants) | 4 | 8 | 2
Participants
  COWS Score <5 | 4 | 7 | 2
  Mild (COWS Score 5-12) | 0 | 1 | 0

17. Primary Outcome: Number of Participants With Clinical Opiate Withdrawal Scale (COWS) at Week 8
Description: as for outcome 7
Time Frame: Week 8
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | PF-06412528 <=20 mg | PF-06412528 >20-40 mg | PF-06412528 >40-80 mg
Number analyzed (Participants) | 4 | 8 | 2
Participants
  COWS Score <5 | 3 | 7 | 1
  Mild (COWS Score 5-12) | 0 | 0 | 1
  Missing | 1 | 1 | 0

18. Primary Outcome: Number of Participants With Clinical Opiate Withdrawal Scale (COWS) at Week 10
Description: as for outcome 7
Time Frame: Week 10
Population: Analysis population: all participants who were screened and received at least 1 dose of PF-06412528 from Week 5-10. Overall number of participants analyzed=0 for arm PF-06412528 >40-80 mg as no participants were evaluable for this outcome measure at Week 10.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-06412528 <=20 mg | PF-06412528 >20-40 mg | PF-06412528 >40-80 mg
Number analyzed (Participants) | 0 | 8 | 0
Participants
  COWS Score <5 |  | 1 |
  Missing |  | 7 |

19. Primary Outcome: Number of Participants With Clinical Opiate Withdrawal Scale (COWS) at Early Termination Before Week 10
Description: as for outcome 7
Time Frame: Early Termination before Week 10 (anytime between Week 5 to Week 10)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | PF-06412528 <=20 mg | PF-06412528 >20-40 mg | PF-06412528 >40-80 mg
Number analyzed (Participants) | 4 | 8 | 2
Participants
  COWS Score <5 | 3 | 6 | 1
  Mild (COWS Score 5-12) | 0 | 1 | 1
  Missing | 1 | 1 | 0

20. Primary Outcome: Apparent Oral Clearance (CL/F) of PF-06412528
Description: Clearance of a drug is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes.
Time Frame: Anytime post-dose on Visit 4 (Week 4)
Population: Data for this outcome measure was not collected, as there were insufficient pharmacokinetic samples due to early termination of the study by the sponsor.
Arm/Group | PF-06412528 <=20 mg | PF-06412528 >20-40 mg | PF-06412528 >40-80 mg
Number analyzed (Participants) | 0 | 0 | 0

21. Primary Outcome: Average Concentration at Steady-state (Css, av) of PF-06412528
Description: Css, av was defines as the average steady state concentration of a drug ("steady state" has been achieved when the rate of drug administration and the rate of drug elimination are equal).
Time Frame: Anytime post-dose on Visit 4 (Week 4)
Population: as for outcome 20
Arm/Group | PF-06412528 <=20 mg | PF-06412528 >20-40 mg | PF-06412528 >40-80 mg
Number analyzed (Participants) | 0 | 0 | 0

22. Secondary Outcome: Number of Participants With Pre-defined Criteria of Vital Signs
Description: Pre-defined criteria of vital signs included supine diastolic blood pressure (DBP) change from baseline greater than or equal to (>=) 20 millimeter of mercury (mmHg): increase and decrease; supine systolic blood pressure (SBP) change from baseline >=30 mmHg: increase and decrease.
Time Frame: Week 1 up to Week 10
Population: Analysis population included all participants who were screened and had received at least 1 dose of PF-06412528 in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-06412528 <=20 mg | PF-06412528 >20-40 mg | PF-06412528 >40-80 mg
Number analyzed (Participants) | 6 | 10 | 3
Participants
  Supine DBP: Change >= 20 mmHg increase | 0 | 2 | 0
  Supine DBP: Change >= 20 mmHg decrease | 1 | 1 | 1
  Supine SBP: Change >= 30mmHg increase | 1 | 0 | 0
  Supine SBP: Change >= 30 mmHg decrease | 0 | 0 | 0

23. Secondary Outcome: Number of Participants With Laboratory Test Abnormalities
Description: Laboratory parameters included: hematology (hemoglobin: <0.8*LLN, hematocrit: <0.8*LLN, red blood cell: <0.8* LLN, platelet <0.5*LLN; >1.75*ULN and white blood cell count <0.6*LLN, neutrophils <0.8* LLN, eosinophils >1.2*ULN, monocytes >1.2*ULN, basophils >1.2*ULN and lymphocytes <0.8* LLN), chemistry (blood urea nitrogen >1.3*ULN, creatinine>1.3*ULN, sodium <0.95*LLN, potassium <0.9*LLN, >1.1*ULN, aspartate aminotransferase >3.0*ULN, alanine aminotransferase >3.0*ULN, total bilirubin >1.5*ULN, alkaline phosphatase >3.0*ULN, albumin <0.8*LLN, total protein<0.8*LLN, >1.2*ULN, Albumin <0.8*LLN, Blood Urea Nitrogen >1.3*ULN, Creatinine >1.3*ULN, HDL Cholesterol <0.8*LLN, Chloride <0.9*LLN, Phosphate <0.8*LLN, Bicarbonate <0.9*LLN, Glucose <0.6*LLN, Creatine Kinase >2.0*ULN, Urobilinogen >=1) and urinalysis (specific gravity <1.003, pH <4.5 urine glucose >=1, ketones >=1 urine protein >=1, urine bilirubin >=1, nitrite >=1, urine leukocytes >=20).
Time Frame: Week 1 up to Week 10
Population: Analysis population included all participants who were screened and had received at least 1 dose of PF-06412528 in the study and evaluated for laboratory abnormalities.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-06412528 <=20 mg | PF-06412528 >20-40 mg | PF-06412528 >40-80 mg
Number analyzed (Participants) | 6 | 8 | 3
Participants | 3 | 7 | 3

24. Secondary Outcome: Apparent Volume of Distribution (Vz/F) of PF-06412528
Description: Volume of distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired plasma concentration of a drug. Apparent volume of distribution after oral dose (Vz/F) is influenced by the fraction absorbed.
Time Frame: Anytime post-dose on Visit 4 (Week 4)
Population: as for outcome 20
Arm/Group | PF-06412528 <=20 mg | PF-06412528 >20-40 mg | PF-06412528 >40-80 mg
Number analyzed (Participants) | 0 | 0 | 0

25. Secondary Outcome: Dose-Exposure Relationship of Metabolites of Morphine, Naltrexone and 6-β-Naltrexol
Time Frame: Anytime post-dose on Visit 4 (Week 4)
Population: as for outcome 20
Arm/Group | PF-06412528 <=20 mg | PF-06412528 >20-40 mg | PF-06412528 >40-80 mg
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Week 1 up to Week 11 (including 1 week of follow-up)
Description: Same event may appear as both an AE and SAE. However, what is presented are distinct events. An event may be categorized as serious in 1 participant and as non-serious in another, or a participant may have experienced both a serious and non-serious event. The study was terminated early therefore the number of participants is small and safety data (all-cause mortality, SAE and other AEs) are presented by dose group.
Arm/Group | PF-06412528 <=20 mg | PF-06412528 >20-40 mg | PF-06412528 >40-80 mg
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/10 | 0/3
Serious Adverse Events (participants affected / at risk) | 2/6 | 2/10 | 2/3
Other Adverse Events (participants affected / at risk) | 5/6 | 9/10 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PF-06412528 <=20 mg (N=6) | PF-06412528 >20-40 mg (N=10) | PF-06412528 >40-80 mg (N=3)
Sickle cell anaemia with crisis (Blood and lymphatic system disorders) | 0 | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0 | 0
Osteomyelitis (Infections and infestations) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1
Bone infarction (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PF-06412528 <=20 mg (N=6) | PF-06412528 >20-40 mg (N=10) | PF-06412528 >40-80 mg (N=3)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1 | 0
Sickle cell anaemia with crisis (Blood and lymphatic system disorders) | 0 | 1 | 0
Palpitations (Cardiac disorders) | 0 | 1 | 0
Ocular hyperaemia (Eye disorders) | 0 | 1 | 0
Visual impairment (Eye disorders) | 0 | 1 | 0
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 0 | 0
Abdominal pain lower (Gastrointestinal disorders) | 1 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 2 | 0
Constipation (Gastrointestinal disorders) | 2 | 2 | 0
Dental caries (Gastrointestinal disorders) | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 3 | 2 | 2
Toothache (Gastrointestinal disorders) | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 2 | 0 | 1
Asthenia (General disorders) | 0 | 0 | 2
Breakthrough pain (General disorders) | 0 | 1 | 0
Chest pain (General disorders) | 1 | 1 | 1
Fatigue (General disorders) | 0 | 1 | 1
Feeling abnormal (General disorders) | 0 | 1 | 0
Feeling cold (General disorders) | 0 | 0 | 1
Mucosal disorder (General disorders) | 0 | 1 | 0
Oedema peripheral (General disorders) | 0 | 1 | 0
Pain (General disorders) | 1 | 1 | 2
Peripheral swelling (General disorders) | 0 | 1 | 1
Pyrexia (General disorders) | 0 | 0 | 1
Ulcer (General disorders) | 0 | 1 | 0
Biliary colic (Hepatobiliary disorders) | 1 | 0 | 0
Cystitis (Infections and infestations) | 0 | 1 | 0
Staphylococcal infection (Infections and infestations) | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 1
Ligament sprain (Injury, poisoning and procedural complications) | 1 | 0 | 0
Penis injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Breath sounds abnormal (Investigations) | 0 | 1 | 0
Lymph node palpable (Investigations) | 0 | 1 | 0
Protein total abnormal (Investigations) | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 2 | 2
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 2 | 1
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 | 0 | 1
Dizziness (Nervous system disorders) | 1 | 1 | 1
Headache (Nervous system disorders) | 3 | 4 | 1
Hypoaesthesia (Nervous system disorders) | 1 | 1 | 1
Hyporeflexia (Nervous system disorders) | 0 | 0 | 1
Migraine (Nervous system disorders) | 0 | 1 | 1
Neuropathy peripheral (Nervous system disorders) | 0 | 1 | 0
Sedation (Nervous system disorders) | 1 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 1
Tension headache (Nervous system disorders) | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 1 | 0
Irritability (Psychiatric disorders) | 0 | 1 | 0
Chromaturia (Renal and urinary disorders) | 0 | 0 | 1
Dysuria (Renal and urinary disorders) | 1 | 1 | 0
Balanoposthitis (Reproductive system and breast disorders) | 0 | 1 | 0
Breast swelling (Reproductive system and breast disorders) | 0 | 1 | 0
Breast tenderness (Reproductive system and breast disorders) | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Nasal ulcer (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Pulmonary pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 2 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 2 | 1
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0

LIMITATIONS AND CAVEATS:
Data for pharmacokinetic outcome measures was not collected, as there were insufficient pharmacokinetic samples due to early termination of the study by the sponsor.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2015-05-26): https://cdn.clinicaltrials.gov/large-docs/54/NCT02101554/Prot_000.pdf
  • Statistical Analysis Plan (2013-12-13): https://cdn.clinicaltrials.gov/large-docs/54/NCT02101554/SAP_001.pdf